CLINICAL TRIAL: NCT00095836
Title: A Phase II Study of ZD 1839 (IRESSA®) in Patients With Advanced Thyroid Cancer
Brief Title: Gefitinib in Treating Patients With Locally Advanced or Metastatic Thyroid Cancer That Did Not Respond to Iodine Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, John Ross Clark, Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-220; P30CA006516 (NIH); ZENECA-IRUSIRES0165 (Other: AstraZeneca); CDR0000393510 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: recurrent thyroid cancer; stage III follicular thyroid cancer; stage III papillary thyroid cancer; stage IV follicular thyroid cancer; stage IV papillary thyroid cancer; anaplastic thyroid cancer; thyroid gland medullary carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Thyroid Carcinoma, Anaplastic; Carcinoma, Medullary | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gefitinib 250mg (Experimental)
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Taken orally once a day for duration of benefit. Treatment is continuous until there is evidence of disease progression or unacceptable toxicity.
  Other Names: ZD1839; IRESSA

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: Phase II trial to study the effectiveness of gefitinib in treating patients who have locally advanced or metastatic thyroid cancer that did not respond to iodine therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the all-measurable-disease response rate in patients with iodine-refractory locally advanced or metastatic thyroid cancer treated with gefitinib.

Secondary

* Determine the toxicity of this drug in these patients.
* Determine progression-free and overall survival of patients treated with this drug.

OUTLINE: This is an open-label study.

Patients receive oral gefitinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed thyroid cancer, metastatic or locally advanced, not amenable or refractory to local therapy and/or radioactive iodine, depending on the cell type.
2. Thyroid cancer that is unresponsive or refractory to radioactive iodine. All medullary and anaplastic thyroid carcinomas will be considered unresponsive on the basis of histopathologic diagnosis alone. Well-differentiated thyroid cancers (papillary and follicular) will be considered refractory if either there is no evidence of uptake on radioactive iodine scanning or tumor growth persists in spite of treatment with radioactive iodine.
3. Measurable disease.
4. Patient is at least 18 years of age.
5. Eastern Cooperative Oncology Group performance status of 0-2.
6. If female and of reproductive potential, a negative β-HCG (human chorionic gonadotropin) and use of effective birth control for the course of the study.
7. Patient is capable of providing signed, informed consent.

Exclusion Criteria:

1. Concurrent chemotherapy, concurrent systemic anticancer treatment, or concurrent radiation therapy. Patients will not be excluded from the study on the basis of prior radiation therapy.
2. Treatment with a non-approved or investigational drug within 30 days before Day 1 of trial treatment.
3. Currently pregnant or nursing.
4. Absolute neutrophil count <1.5 × 109/L, platelet count < 75 × 109/L, bilirubin > 1.5 × normal, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × normal.
5. Serum creatinine greater than Common Toxicity Criteria (CTC) grade 2.
6. Concomitant use of phenytoin, carbamazepine, barbiturates, rifampin, St John's Wort.
7. Concomitant use of systemic retinoids, cyclosporine, verapamil, diltiazem, nicardipine, nifedipine, nitrendipine, erythromycin, theophylline, ketoconazole, itraconazole, and antihistamines such as terfenadine and astemizole.
8. Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy.
9. Incomplete healing from previous oncologic or other major surgery.
10. Known severe hypersensitivity to ZD1839 or any of the excipients of this product.
11. As judged by the investigator, any evidence of severe or uncontrolled systemic disease

    (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
12. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial.
13. Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-03 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Clark, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Pennell NA, Daniels GH, Haddad RI, Ross DS, Evans T, Wirth LJ, Fidias PH, Temel JS, Gurubhagavatula S, Heist RS, Clark JR, Lynch TJ. A phase II study of gefitinib in patients with advanced thyroid cancer. Thyroid. 2008 Mar;18(3):317-23. doi: 10.1089/thy.2007.0120. PMID 17985985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from Massachusetts General Hospital and the Dana-Farber Cancer Institute
Period: Overall Study
Arm/Group | Gefitinib 250mg
Started | 27
Completed | 23
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gefitinib 250mg
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status.
  0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  1. - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  2. - Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours)
  Participants
    0-1 | 25
    2 | 2
Stage [Count of Participants; unit: Participants]
  Locally Advanced | 2
  Metastatic | 25
Metastatic sites [Count of Participants; unit: Participants] — Population: Participants with metastatic cancer
  Participants
    Lung-only: number analyzed (Participants) | 25
    Lung-only | 10
    Lung + extra-pulmonary metastases: number analyzed (Participants) | 25
    Lung + extra-pulmonary metastases | 15
Prior therapy [Number; unit: participants]
  Radioactive iodine | 17
  Chemotherapy | 6
  External beam radiotherapy | 23
Histology [Count of Participants; unit: Participants]
  Papillary | 11
  Follicular | 6
  Anaplastic | 5
  Medullary | 4
  Hürthle cell | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate at 3, 6, and 12 Months
Description: Response rate as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Tumor assessment is performed within 4 weeks of initiation of treatment and then every 8 weeks. If a patient has stable disease for four tumor assessments (6 months), then tumor assessment may occur every 4 months. If the patient continues to experience stable disease after 2 years, tumor assessments may occur every 6 months. If the patient continues to experience stable disease after 5 years, tumor assessments may occur once a year.
  Complete Response (CR): Disappearance of all target lesions
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
Time Frame: 3 Months, 6 Months, 1 Year
Population: Two patients lost to follow-up prior to assessment of tumor response
Measure: Number; unit: participants
Arm/Group | Gefitinib 250mg
Number analyzed (Participants) | 25
participants
  Complete Response : 3 Months | 0
  Partial Response : 3 Months | 0
  Stable Disease : 3 Months | 12
  Progressive Disease : 3 Months | 13
  Complete Response : 6 Months | 0
  Partial Response : 6 Months | 0
  Stable Disease : 6 Months | 6
  Progressive Disease : 6 Months | 19
  Complete Response : 12 Months | 0
  Partial Response : 12 Months | 0
  Stable Disease : 12 Months | 3
  Progressive Disease : 12 Months | 22

2. Secondary Outcome: Toxicity
Description: Drug related toxicity as assessed by NCI CTCAE that occurred in more than 10% of patients
Time Frame: Through study completion, on average 12 months
Measure: Number; unit: participants
Arm/Group | Gefitinib 250mg
Number analyzed (Participants) | 27
participants
  Rash: Grade 0 | 13
  Rash: Grade 1 | 9
  Rash: Grade 2 | 3
  Rash: Grade 3 | 2
  Diarrhea: Grade 0 | 16
  Diarrhea: Grade 1 | 8
  Diarrhea: Grade 2 | 2
  Diarrhea: Grade 3 | 1
  Nausea: Grade 0 | 22
  Nausea: Grade 1 | 5
  Anorexia: Grade 0 | 24
  Anorexia: Grade 1 | 3

3. Secondary Outcome: Median Progression-free Survival
Description: The median progression-free survival as assessed by RECIST criteria (Response Evaluation Criteria In Solid Tumors) measured from the time of enrollment until disease progression or death.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or the appearance of new lesions.
Time Frame: From the time of enrollment until disease progression or death, whichever came first
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib 250mg
Number analyzed (Participants) | 27
Months | 3.7 [1.8 to 5.7]

4. Secondary Outcome: Overall Survival
Description: The median overall survival time, measured from the time of enrollment until death.
Time Frame: 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Gefitinib 250mg
Number analyzed (Participants) | 27
Months | 17.5 [9.2 to NA] — Participant was still alive at time of assessment

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1.5 years
Description: During routine visits subjects will be assessed for toxicity using physical examination and laboratory tests. Assessments are performed every 4 weeks while on treatment. If a participant has experienced no grade 3 or 4 toxicity for a 6-month time period, toxicity may be assessed every 2 months. If If the patient continues to do well after 2 years, assessment may be extended to every 3 months.
Arm/Group | Gefitinib 250mg
All-Cause Mortality (participants affected / at risk) | 2/27
Serious Adverse Events (participants affected / at risk) | 6/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib 250mg (N=27)
Hematuria (Renal and urinary disorders) | 1 (1)
Airway obstruction (mucous) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdomen- pain (Gastrointestinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib 250mg (N=27)
Hemoglobin (Blood and lymphatic system disorders) | 4 (27)
Hypotension (Vascular disorders) | 4 (66)
Fatigue (General disorders) | 11 (49)
Fever w/o neutropenia (General disorders) | 2 (5)
Insomnia (General disorders) | 2 (8)
Odor (patient odor) (General disorders) | 4 (22)
Constitutional, other (General disorders) | 2 (6)
Bruising (Skin and subcutaneous tissue disorders) | 6 (57)
Induration/fibrosis (Skin and subcutaneous tissue disorders) | 2 (4)
Photosensitivity (Skin and subcutaneous tissue disorders) | 15 (110)
Skin-other (Skin and subcutaneous tissue disorders) | 4 (8)
Anorexia (Gastrointestinal disorders) | 6 (27)
Constipation (Gastrointestinal disorders) | 3 (39)
Teeth development (Gastrointestinal disorders) | 3 (40)
Fistula, Duodenum (Gastrointestinal disorders) | 4 (26)
Fistula, Gallbladder (Gastrointestinal disorders) | 6 (45)
Fistula, Pharynx (Gastrointestinal disorders) | 2 (2)
Fistula, Stomach (Gastrointestinal disorders) | 11 (66)
Colon, hemorrhage (Gastrointestinal disorders) | 2 (28)
Infection w/ gr3-4 neut, appendix (Infections and infestations) | 2 (2)
Confusion (Nervous system disorders) | 2 (14)
Extrapyramidal movement (Nervous system disorders) | 2 (3)
Laryngeal nerve dysfunction (Nervous system disorders) | 2 (21)
Leak, CSF (Nervous system disorders) | 2 (7)
Leukoencephalopathy (Nervous system disorders) | 2 (7)
Mental status (Nervous system disorders) | 2 (30)
Anxiety (Nervous system disorders) | 4 (34)
Ocular-other (Eye disorders) | 2 (2)
Back, pain (Musculoskeletal and connective tissue disorders) | 6 (39)
Bladder, pain (Renal and urinary disorders) | 2 (3)
Pain-other (General disorders) | 8 (28)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 9 (99)
(DLCO) (Respiratory, thoracic and mediastinal disorders) | 6 (37)
Fistula lung (Respiratory, thoracic and mediastinal disorders) | 2 (38)
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal/GU-other (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes